CLINICAL TRIAL: NCT04069624
Title: Kentucky Women's Justice Community Opioid Innovation Network
Acronym: W-JCOIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michele Staton (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Michele Staton, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 51656; 1UG1DA050069 (NIH)
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Opioid-use Disorder
Keywords: MOUD; OUD; Telehealth; Navigator
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Services as Usual (SAU) (Active Comparator): Substance abuse program (SAP) managed by the Kentucky Department of Corrections, with the option to initiate MOUD prior to jail release.
  Interventions: Other: Services as Usual
- MOUD Pre-Treatment Telehealth (Experimental): Telehealth connection to a community MOUD provider.
  Interventions: Behavioral: MOUD Pre-Treatment Telehealth
- MOUD Pre-Treatment Telehealth and Peer Navigator (Experimental): Telehealth connection to a community MOUD provider, in addition to a peer navigator
  Interventions: Behavioral: MOUD Pre-Treatment Telehealth and Peer Navigator

INTERVENTIONS:
Behavioral: MOUD Pre-Treatment Telehealth — Opioid use disorder (OUD) assessment, medical evaluation, and medications to treat opioid use disorder (MOUD) education with a MOUD provider during incarceration via telehealth
  Arms: MOUD Pre-Treatment Telehealth
Behavioral: MOUD Pre-Treatment Telehealth and Peer Navigator — Opioid use disorder (OUD) assessment, medical evaluation, and medications to treat opioid use disorder (MOUD) education with a MOUD provider during incarceration via telehealth. Additionally, participants will be connected with a Peer Navigator who will meet with them via telehealth prior to release and provide ongoing support by telephone post-release.
  Arms: MOUD Pre-Treatment Telehealth and Peer Navigator
Other: Services as Usual — Medications to treat opioid use disorder (MOUD) pre-treatment.
  Arms: Services as Usual (SAU)

SUMMARY:
This trial will test the effectiveness of delivering medication for opioid use disorder (MOUD) pre-treatment via telehealth, alone and with peer navigation, to increase MOUD initiation and maintenance in the community following jail release. This trial will focus on incarcerated women in 6 experimental and 3 control sites in Kentucky. Enrollment is not open to the general public.

DETAILED DESCRIPTION:
This study will incorporate random assignment for two study conditions: medication for opioid use disorder (MOUD) PreTreatment Telehealth or MOUD PreTreatment Telehealth with Peer Navigation using a rigorous randomized block design. Women in the experimental conditions will be stratified by sites (6 sites; 3 urban and 3 non-urban) and by offender classification level of felony versus misdemeanor (due to potential differences in community supervision). Three comparison sites with existing jail-based MOUD treatment for women will not be randomized but will be included in analyses within planned, non-randomized comparisons.

1. MOUD PreTreatment Telehealth: Participants who screen positive for moderate to high-risk opioid use and complete the baseline interview will be connected via telehealth to the community MOUD provider for a psychosocial assessment. The study data coordinator will assist with linking the participant to the community MOUD provider via telehealth, as well as collecting initial in-person biological specimens for medical evaluation. The psychosocial assessment with the community MOUD provider will involve a more detailed examination of OUD using the Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 criteria. Type of medication (naltrexone, buprenorphine, or methadone) will depend on the psychosocial assessment and medical evaluation. Indications for the most appropriate course of treatment will be determined by the community MOUD provider in conjunction with the study participant. Women in this condition will also receive general education about MOUD options including risks and benefits, and they will be given the opportunity to ask questions about the medication. The community MOUD provider will also use motivational interviewing to assess each woman's readiness to engage in MOUD and to better understand possible barriers to MOUD utilization. At the end of the education session, the study participant and the MOUD community provider will develop a re-entry plan for ongoing care, which will include a plan for insurance coverage of medications in the community.
2. MOUD PreTreatment Telehealth + Peer Navigation: In addition to MOUD PreTreatment Telehealth, women in this arm will be connected with a peer, a woman in recovery who is employed by Voices of Hope (VOH) in Lexington, KY. Peer Navigators will be located in Lexington through a partnership with VOH. VOH is a non-profit recovery support organization which provides peer recovery support services. In conjunction with the study data coordinators, the Peer Navigator will schedule an initial session via telehealth with the participant, assist with scheduling a follow-up appointment with the community MOUD provider, and provide recovery support for community MOUD initiation and maintenance. Peer Navigators will be certified Peer Support Specialists trained and supervised by VOH in accordance with state statutory requirements. When a woman returns to the community, Peer Navigators will engage her in weekly telephone recovery services (TRS) for 12 weeks, which may include identifying personal goals and strength-based, practical strategies for success. In addition to MOUD linkages to care, Peer Navigators will suggest strategies to maintain sobriety and improve recovery capital, including safe housing, transportation, financial counseling, continued education, employment skills, and sober social activities.
3. Services as Usual: Women in this arm will not be randomized, but will receive substance abuse treatment as usual in three comparison jail sites. Each of these jails has a women's substance abuse program (SAP) managed by the Kentucky Department of Corrections (KY-DOC with the option to initiate MOUD prior to jail release. These programs operate as modified therapeutic communities with transitional support following release.

ELIGIBILITY:
Inclusion Criteria:

* ASSIST opioid (prescription or street) score of 4+
* Willingness to participate in MOUD pre-treatment
* Incarceration period of at least 7 days

Exclusion Criteria

• Cognitive impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The number of participants who initiate MOUD | 13 months
  Any initiation of MOUD post-release over the study period

SECONDARY OUTCOMES:
Medication Type | 13 months
  Percentage of participants on naltrexone, buprenorphine or methadone.
Opioid Relapse | 13 months
  Percentage of participants relapsing, measured by self-report or drug screen.
Treatment Retention | 13 months
  Length of time in treatment
Recidivism | 12 months
  Percent of participants returning to custody
Overdose Rates | 13 months
  Percentage of participants who overdose (medical attention needed for revival)
Criminal Activity | 12 months
  Percent of participants engaging in criminal activity (self-report or arrest records)

OTHER OUTCOMES:
Total Annual Intervention Cost | 5 years
  Total annual intervention cost
Average Participant Cost | 13 months
  Average intervention cost per participant
Incremental Cost-Effectiveness Ratio | 5 years
  Cost per unit outcome of interventions versus services as usual
Public Health Cost of Opioid Relapse | 5 years
  Cumulative estimated cost of hospitalizations, treatments, loss of work, child welfare, and other services related to relapse.
Public Safety Cost of Recidivism and Criminal Activity | 5 years
  Cumulative estimated cost of return to custody, arrests, and other social costs of recidivism.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Staton, MSW, PhD, Principal Investigator — University of Kentucky
Locations (9):
- United States (9):
  - Hardin County Detention Center, Elizabethtown, Kentucky
  - Harlan County Detention Center, Harlan, Kentucky
  - Henderson County Detention Center, Henderson, Kentucky
  - Marion County Detention Center, Lebanon, Kentucky
  - Grayson County Detention Center, Leitchfield, Kentucky
  - Laurel County Correctional Center, London, Kentucky
  - Pike County Detention Center, Pikeville, Kentucky
  - Shelby County Detention Center, Shelbyville, Kentucky
  - Grant County Detention Center, Williamstown, Kentucky

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data at this time.

REFERENCES:
- [Derived] Staton M, Levi M, Winston E, B Oser C, Fallin-Bennett A, Dickson M, Matthew Webster J, Leukefeld C, Tillson M. Examining use of telehealth in jails: linking women to community OUD services. BMC Womens Health. 2024 Oct 4;24(1):549. doi: 10.1186/s12905-024-03394-4. PMID 39367439